CLINICAL TRIAL: NCT05279313
Title: A Phase 3, Multicenter, Open-label, Long-term Trial Evaluating the Long-term Safety and Tolerability of Once Daily Centanafadine Capsules in Children and Adolescents (4 to 17 Years of Age, Inclusive) With Attention-deficit/Hyperactivity Disorder (ADHD).
Brief Title: A Trial of Centanafadine Long-term Safety in Children and Adolescents With Attention-deficit/Hyperactivity Disorder.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00017
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Centanafadine; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Centanafadine Hydrochloride (Experimental): * Adolescents (13 to 17 years of age, inclusive) to receive 328.8 mg daily.
  * Children (4 to 12 years of age, inclusive) will receive weight-based doses of centanafadine ranging from 82.2 mg to 328.8 mg daily
  Interventions: Drug: Centanafadine Hydrochloride

INTERVENTIONS:
Drug: Centanafadine Hydrochloride — Capsule
  Other Names: Centanafadine; Centanafadine XR; EB-1020

SUMMARY:
To evaluate long-term safety exposure

DETAILED DESCRIPTION:
This open-label study will assess the overall safety and tolerability of centanafadine once daily extended-release capsules in pediatric subjects (ages 4-17 years). The study will accept rollover subjects from double-blind parent trials and individuals that did not participate in one of the double-blind parent trials, may enroll as De Novo subjects after meeting all required study entry criteria. All subjects will complete a minimum of 52 weeks and may continue until all enrolled subjects within the age group the subject was in at the start of their participation in the trial (13 to 17 years; 6 to 12 years; 4 to 5 years) have had a chance to reach the Week 52 visit.

ELIGIBILITY:
Rollover subjects from double-blind parent trials inclusion criteria:

* Subjects who completed the 6-week double-blind treatment period and the 7 (+2) day follow-up in a double-blind parent trial and who, in the opinion of the investigator, could potentially benefit from centanafadine QD XR for ADHD

De novo subjects inclusion criteria:

* Males and females aged 4 to 17 years (inclusive) at the time of informed consent/assent.
* A primary diagnosis of ADHD based on DSM-5 diagnosis criteria as confirmed with the MINI KID.
* A minimum symptoms total raw score of ≥ 28 on the ADHD-RS-5 at baseline.
* A score of 4 or higher on the CGI-S-ADHD at baseline.
* Subjects aged 4 or 5 years only; has failed adequate psychotherapy or in the investigator's opinion, is severe enough to require pharmacotherapy in the absence of prior psychotherapy.

Rollover subjects from double-blind parent trials exclusion criteria:

* Subjects who, during the double-blind parent trials, experienced, in the opinion of the investigator, poor tolerability to IMP or whose safety assessments resulted in new concerns that would suggest the subject may not be appropriate for a 52-week treatment with IMP.

De novo subjects exclusion criteria:

* A comorbid diagnosis of: Tourette's Disorder, Generalized Anxiety Disorder that is severe enough to interfere with trial procedures, Panic Disorder, Conduct Disorder, Psychosis, Post-traumatic Stress Disorder, Bipolar Disorder, Autism Spectrum Disorder, Binge Eating Disorder (adolescents only), Anorexia (adolescents only), Bulimia (adolescents only), Oppositional Defiant Disorder that is severe enough to interfere with trial conduct (allowed if it is not the primary focus of treatment), Obsessive-Compulsive Disorder that is severe enough to interfere with trial conduct (allowed if it is not the primary focus of treatment), MDD with current major depressive episode, or has required treatment within the 3 months prior to screening, or in investigator's opinion, MDD may worsen or could be expected to require treatment during the course of this trial.
* Subjects who are breast-feeding and/or have a positive pregnancy test result prior to receiving IMP.
* A significant risk of committing suicide based on history and the investigator's clinical judgment, or routine psychiatric status examination, current suicidal behavior, Imminent risk of injury to self, active suicidal ideation, history of suicidal behavior (over the last 6 months).
* Body weight < 13 kg
* BMI ≥ 40 kg/m2
* Has initiated, changed, or discontinued receiving psychological interventions for ADHD within the 30 days before the screening visit, or are anticipated to start new treatment during the trial.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 680 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs) will be assessed to determine long-term safety and tolerability of Centanafadine QD XR Capsules. | Minimum duration of 52 weeks, up to a maximum of approximately 136 weeks or early termination.

CONTACTS AND LOCATIONS:
Locations (85):
- United States (83):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - The Center for Clinical Trials, Inc., Saraland, Alabama
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Care Access, Beverly Hills, California
  - Proscience Research Group, Culver City, California
  - Sun Valley Research Center, Inc., Imperial, California
  - Long Beach Clinical Trials Services, Inc, Long Beach, California
  - NRC Research Institute, Orange, California
  - SDS Clinical Trials Inc, Santa Ana, California
  - CMB Clinical Trials, Santee, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Mindscapes Counseling LLC DBA Comprehensive Psychiatric Care, PC, Norwich, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - West Broward Outpatient Site, Lauderhill, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Clinical Trials Solution, Miami, Florida
  - Care Research Inc, Miami, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - ABRI, Miami, Florida
  - Ivetmar Medical Group, LLC, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Anchor Medical Research, LLC, Miami, Florida
  - RM Medical Research, Inc., Miami Lakes, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Apg Research, Llc, Orlando, Florida
  - Space Coast Neuropsychiatric Research Institute, Palm Bay, Florida
  - University of South Florida, Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - CenExcel-iResearch, LLC, Decatur, Georgia
  - Velocity Clinical Research Boise, Meridian, Idaho
  - American Medical Research, Inc., Chicago, Illinois
  - AMR-Baber Research Inc, Naperville, Illinois
  - Qualmedica Research, Evansville, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Qualmedica Research LLC, Bowling Green, Kentucky
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Sisu BHR, LLC, Springfield, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - St. Charles Psychiatric Associates / Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Vector Clinical Trials, Las Vegas, Nevada
  - Albuquerque Neuroscience, INC, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - Onsite Clinical Solutions LLC, Charlotte, North Carolina
  - University of Cincinnati Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cincy Science, West Chester, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Paradigm Research Professionals LLC, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - Inquest Clinical Research Baytown Health LLC, Baytown, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Javara Inc., Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Allure Health at Mt. Olympus Medical Research, Friendswood, Texas
  - Synergy Groups Medical LLC, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - AIM Trials, LLC, Plano, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Velocity Clinical Research Salt Lake City, West Jordan, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Inc. dba Core Clinical Research, Everett, Washington
- Center for Pediatric Excellence, Ottawa, Ontario, Canada
- Barbara Diaz Hernandez MD Research, Inc., San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com